CLINICAL TRIAL: NCT07384000
Title: The Efficacy of Single Puncture Technique of Rectus Sheath Block Combined With Transversus Abdominis Plane Block Versus External Oblique Intercostal Plane Block for Pain Control After Laparoscopic Cholecystectomy.
Brief Title: Comparison Between External Oblique Intercostal Plane Block and Rectus Sheath Block Combined With Transversus Abdominis Plane Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Osama Mohamed Hassan, Principal investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: nerve block in pain management
Record Dates: First submitted 2026-01-11; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Pain Management; Anesthesia , Analgesia; Nerve Block
Keywords: Comparison Between External Oblique Intercostal Plane Block and Rectus Sheath Block Combined With Transversus Abdominis Plane Block
MeSH Terms: conditions — Agnosia | interventions — Control Groups; Nalbuphine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in parallel to one of three groups: (1) external intercostal plane block, or (2) combined rectus sheath block and transversus abdominis plane block by single puncture technique (3) the control group recieve nalbuphine . Each participant receives only one intervention according to group allocation.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- external intercostal plane block intervention with ultra sound (Active Comparator): Patients in this group will receive (EOIPB) bilaterally, the block will be performed under ultrasound guidance after induction of general anesthesia using 20 ml of 0.25% bupivacaine injected into the external oblique intercostal plane on each side.
  Interventions: Procedure: External intercostal plane puncture
- single-puncture technique of (RSB) combined with (TAPB) by ultra sound (Active Comparator): Patients in this group will receive rectus sheath block (RSB) combined with transversus abdominis plane block (TAPB) bilaterally via single puncture, the block will be performed under ultrasound guidance after induction of general anesthesia using 20 ml of 0.25% bupivacaine divided into 10 ml of 0.25% bupivacaine will be injected when the needle reaches the posterior rectus abdominis sheath and pierces the anterior layer of the posterior sheath, Then, the needle will break through the posterior layer of the tendon to the transversus abdominis plane and another 10 ml of 0.25% bupivacaine will be injected into transversus abdominis plane .
  Interventions: Procedure: the single-puncture technique of (rectus sheath block) combined with (Transversus abdominis plane block)
- control group (nalbuphine) (Placebo Comparator): Patients in this group will not receive any intervention or nerve block.
  Interventions: Drug: control group (nalbuphine)

INTERVENTIONS:
Procedure: External intercostal plane puncture — Patients in this group will receive external intercostal plane block bilaterally, the block will be performed under ultrasound guidance after induction of general anesthesia using 20 ml of 0.25% bupivacaine injected into the external oblique intercostal plane on each side.
  Arms: external intercostal plane block intervention with ultra sound
Drug: control group (nalbuphine) — Patients in this group will not receive any intervention or nerve block.
  Arms: control group (nalbuphine)
Procedure: the single-puncture technique of (rectus sheath block) combined with (Transversus abdominis plane block) — Patients in this group will receive rectus sheath block (RSB) combined with transversus abdominis plane block (TAPB) bilaterally via single puncture, the block will be performed under ultrasound guidance after induction of general anesthesia using 20 ml of 0.25% bupivacaine divided into 10 ml of 0.25% bupivacaine will be injected when the needle reaches the posterior rectus abdominis sheath and pierces the anterior layer of the posterior sheath, Then, the needle will break through the posterior layer of the tendon to the transversus abdominis plane and another 10 ml of 0.25% bupivacaine will be injected into transversus abdominis plane .
  Arms: single-puncture technique of (RSB) combined with (TAPB) by ultra sound

SUMMARY:
Effective perioperative pain management remains a cornerstone in enhancing recovery and improving patient outcomes in laparoscopic cholecystectomy. This minimally invasive procedure, although less traumatic compared to open surgery, can still lead to significant postoperative pain, particularly in the early hours following the operation. Insufficient pain control may result in delayed mobilization, prolonged hospital stays, and increased opioid consumption, which are associated with adverse side effects and a heightened risk of complications . Regional anesthesia techniques have garnered significant attention for their ability to provide localized, opioid-sparing analgesia, thereby improving postoperative recovery profiles.External Oblique Intercostal Plane Block (EOIP) is a relatively new regional anesthesia technique targeting the intercostal nerves (T7-T11) as they traverse the plane between the external and internal oblique muscles. This block has demonstrated efficacy in controlling postoperative pain for upper abdominal surgeries, including laparoscopic cholecystectomy. By selectively anesthetizing the sensory branches of the thoracoabdominal nerves, the EOIP block provides localized analgesia with minimal motor blockade, making it an ideal choice for early mobilization (Ouchi et al., 2020).Recent advancements in ultrasound-guided techniques have improved the precision and safety of the EOIP block, allowing for consistent blockade of the targeted nerves. Clinical trials have highlighted its ability to reduce the pain significantly in the first 24 hours postoperatively, along with a marked decrease in the need for rescue analgesics. Tranrversus abdominis plane block (TAP) , first described in the early 2000s, has undergone several modifications to improve its efficacy in abdominal surgeries. The subcostal TAP block targets the anterior branches of the lower thoracic nerves (T6-T9) to provide analgesia to the upper abdominal wall. This technique is particularly suited for laparoscopic cholecystectomy, where the pain originates predominantly from the pari0etal peritoneum and abdominal wall incisions.The single puncture technique of Rectus sheath block (RSB) combined with transversus abdominis plane block (TAPB) represents a more streamlined approach to abdominal wall analgesia. ultrasonography (US) guidance for peripheral nerve blocks has become more and more popular. Transversus abdominis plane block (TAPB) and US-guided rectus sheath block (RSB) have been utilized in abdominal surgeries and have shown strong analgesic effects. Prior researches has demonstrated that in abdominal surgery, US-guided (TAPB) in conjunction with (RSB) had superior analgesic effects than either (TAPB) or (RSB) alone. Currently, multipoint nerve block procedures are generally applied in clinical practice, but they are difficult and can increase the patient's suffering. A novel method is proposed based on the neuromuscular anatomy and the location of the incisiopn in laparoscopic upper abdominal surgery: US-guided transverse abdominis plane and rectus sheath block one-puncture .

DETAILED DESCRIPTION:
This study aims to investigate the analgesic efficacy of external oblique intercostal plane (EOIPB) versus single puncture technique of rectus sheath block (RSB) combined with transversus abdominis plane block (TAPB) after laparoscopic cholecystectomy.

Primary Outcome:

The primary outcome of the study will be the amount of opoid (nalbuphine) consumption in the first 24 hours postoperatively.

Secondary Outcomes:

the analgesic efficacy (Sensory assessment) by defined dermal zones in the first 24 hours postoperatively.

pain intensity at rest and during coughing using verbal rating scale in the first 24 hours postoperatively.

Patient satisfaction in the first 24 hours postoperatively. The hemodynamic changes. Time to first rescue analgesia. First off-bed activity Incidence of block-related complications. Signs of local anesthetic toxicity hypotension ,bradycardia ,tachyarrhythmia, postoperative nausea and vomiting (PONV) and dizziness.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic cholecystectomy
* American Society of Anesthesiologists (ASA) 1-II
* aged 18-70 years
* both genders will be included.
* body mass index (BMI) ≤ 35 kg/m2.

Exclusion Criteria:

* coagulation disorders
* liver/kidney disease
* History of abdominal surgery
* infection in the block application area
* chronic opioid use
* local anesthetic (LA) allergy
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Decrase the consumption of opioids | Intraoperative, immediately postoperative , 2 hours post operative , 4 hours post operative , 6 hours postoperative, 12 hours postoperative, 24 hours postoperative
  The primary outcome of the study will be the amount of opoid (nalbuphine) consumption in the first 24 hours postoperatively.

SECONDARY OUTCOMES:
The analgesic efficacy (sensory assessment) | First hour, second hour , sixth hour, 12th hour , 24th hour postoperatively
  Sensory assessment by defined dermal zones at 1, 2, 6, 12, and 24 hours postoperatively.
  The specific dermal zones will be described by vertical lines at the midline (A), mid-clavicular line (B), anterior axillary line (C), mid-axillary line (D), posterior axillary line (E), infrascapular line (F), and back midline (J).
  Four horizontal lines at the xiphoid level (a),12th costal level (b), the umbilical level (c), the anterior superior iliac spine to the pubic symphysis line (d), and extension to the back to the anterior superior iliac spine level (e).
  An additional zone will be defined as the upper 1/3 of the front thigh . Sensory assessment will be achieved using 70% ethyl alcohol swab and pinprick at 1,2, 6, 12, and 24 hours postoperatively after extubation at specific dermal zones divided by anatomic landmark lines on the abdomen, the back, and the thigh.
  Effective analgesic efficacy was defined as loss of cold temperature sensation to alcohol swab or loss of pinprick pain sensat
Pain intensity | Immediately postoperative, 2 hours postoperative, 4 hours postoperatively, 6 hours postoperative, 12 hours postoperative, 24 hours postoperative
  pain intensity will be assessed at rest and during coughing using verbal rating scale (Jensen & Karoly 1992) every hour till 6 hour, then every 2 hours till 12 hours, then every 4 hours till 24 hours. postoperatively as: No pain (=1) , Mild pain(=2)
  , Moderate pain(=3) , Sever pain(=4).
Off bed activity | 24 hours postoperative
  time of the first off-bed activity after surgery in minutes , comparison between all arms and intervention

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yu S, Wen Y, Lin J, Yang J, He Y, Zuo Y. Combined rectus sheath block with transverse abdominis plane block by one puncture for analgesia after laparoscopic upper abdominal surgery: a randomized controlled prospective study. BMC Anesthesiol. 2024 Feb 9;24(1):58. doi: 10.1186/s12871-024-02444-6. PMID: 38336613; PMCID: PMC10854179.
- See also: White L, Ji A. External oblique intercostal plane block for upper abdominal surgery: use in obese patients. Br J Anaesth. 2022 May;128(5):e295-e297. doi: 10.1016/j.bja.2022.02.011. Epub 2022 Mar 3. PMID: 35249704. — https://pubmed.ncbi.nlm.nih.gov/35249704/
- See also: Yu S, Wen Y, Lin J, Yang J, He Y, Zuo Y. Combined rectus sheath block with transverse abdominis plane block by one puncture for analgesia after laparoscopic upper abdominal surgery: a randomized controlled prospective study. BMC Anesthesiol. 2024 Feb 9;2 — https://pubmed.ncbi.nlm.nih.gov/38336613/